CLINICAL TRIAL: NCT06235983
Title: An Open-label, Single-arm, Multicenter, Phase 1 Study to Investigate the Pharmacokinetics, Safety, Tolerability, and Antitumor Activity of LY3537982 in Chinese Patients With KRAS G12C-Mutant Advanced Solid Tumors
Brief Title: A Study of LY3537982 in Chinese Participants With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18737; J3M-MC-JZQC (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Advanced Solid Tumors
Keywords: Pharmacokinetics; Safety and Tolerability; Chinese

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- LY3537982 (Experimental): LY3537982 administered orally.
  Interventions: Drug: LY3537982

INTERVENTIONS:
Drug: LY3537982 — Administered orally.
  Other Names: Olomorasib

SUMMARY:
This is an open-label, single-arm, multicenter, Phase 1 study of LY3537982 as monotherapy in Chinese participants with KRAS G12C-mutant advanced solid tumors. The main purpose of this study is to determine how much of LY3537982 gets into the bloodstream and how long it takes the body to eliminate it in Chinese participants. The safety, tolerability and preliminary efficacy of LY3537982 will also be evaluated. Approximately 12 patients will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* - Native Chinese participants must be of an acceptable age to provide informed consent.
* Have measurable disease per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST version 1.1).
* Have disease with evidence of KRAS G12C mutation
* Have a histologically or cytologically proven diagnosis of locally advanced, unresectable, and/or metastatic cancer and must be appropriate candidates for study treatment.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Have adequate laboratory parameters.
* Must be able to swallow capsules or tablets.
* Estimated life expectancy ≥12 weeks

Exclusion Criteria:

* Have disease suitable for local therapy administered with curative intent.
* Have an active fungal, bacterial, and/or active untreated viral infection,
* Have a serious pre-existing medical condition(s) that would preclude participation in this study.
* Have a serious cardiac condition.
* Have untreated active symptomatic central neural system (CNS) malignancy or metastasis and/or carcinomatous meningitis.
* Have received prior treatment with any KRAS G12C small molecule inhibitor.
* Females who are pregnant or lactating.
* Have a known allergic reaction against any of the components of the study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Maximum Observed Plasma Concentration (Cmax) of LY3537982 | Predose approximately up to 18 weeks
  PK: Cmax of LY3537982
PK: Area Under the Plasma Concentration Versus Time Curve (AUC) of LY3537982 | Predose approximately up to 18 weeks
  PK: AUC of LY3537982

SECONDARY OUTCOMES:
Objective Response Rate (ORR): ORR assessed per Response Evaluation Criteria in Solid Tumors version 1.1 (RESIST v1.1). | First dose on day 1 approximately up to 3 years
  ORR: ORR assessed per Response Evaluation Criteria in Solid Tumors version 1.1 (RESIST v1.1).
Disease control rate (DCR): DCR assessed per Response Evaluation Criteria in Solid Tumors version 1.1 (RESIST v1.1). | First dose on day 1 approximately up to 3 years
  DCR: DCR assessed per Response Evaluation Criteria in Solid Tumors version 1.1 (RESIST v1.1).
Progression-free survival (PFS): PFS assessed per Response Evaluation Criteria in Solid Tumors version 1.1 (RESIST v1.1). | First dose on day 1 approximately up to 3 years
  PFS: PFS assessed per Response Evaluation Criteria in Solid Tumors version 1.1 (RESIST v1.1).

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- China (3):
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No